CLINICAL TRIAL: NCT05613049
Title: Confounding Factors of Chronic Endometritis in Women With Reproductive Failure
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2022.339
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: IVF
Keywords: chronic endometritis; confounding factors; reproductive failure; infertility; IVF; infertility women
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Patient will be invited to do endometrial sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational group: Patients have 2 or more miscarriage or repeated implantation failure (RIF), or infertile women would be invited to do endometrial sampling (ES) procedure. The ES will be conducted randomly or when women undergo hysteroscopy or obtained precisely 7 days after LH surge. It will be obtained using a Pipelle sampler as an outpatient procedure.

INTERVENTIONS:
Other:  — If the CE is high, antibiotics will be given to the patients as usual practice in hospitals.

SUMMARY:
The aim of the study is to investigate the confounding factors of chronic endometritis and therapeutic benefits of antibodies targeting plasma cells in women with reproductive failure.

DETAILED DESCRIPTION:
Eligible women, based on the inclusion and exclusion criteria, will be recruited from the IVF and/ or miscarriage clinic in the Prince of Wales Hospital/ CUHK medical centre (CUMC). Endometrial sampling (ES) will alternatively be conducted during mid-luteal phase. In natural cycles, all the subjects will have a daily urine test from day 9 of the menstrual cycle to identify the Luteinizing Hormone (LH) surge. The ES will be obtained precisely 7 days after LH surge. In artificial cycles, 6mg estradiol will be given daily orally from day 2 of the menstrual cycle for 14+/-1-2 days. Transvaginal ultrasound will be performed on day 14 of the estrogen therapy to assess the endometrial thickness and to exclude ovarian activity. If endometrial thickness is ≥8 mm, plasma progesterone level is < 4nmol/L, progesterone will be commenced using either Endometrin (Ferring, Saint-Prex, Switzerland) 100 mg TDS vaginally. ES will be obtained using a Pipelle sampler as an outpatient procedure. The ES will be obtained precisely 5 days after progesterone supplementation.

Immunohistochemical staining will be used to determine plasma cells by using a mouse antihuman monoclonal primary anti-CD138 antibody and anti-CD38 antibody. The total number of plasma cell present in the stroma of the entire specimen will be determined and expressed as plasma cell count per unit area of the specimen. If CE is present, antibiotics will be given following the guideline from the Hospital Authority (HA). Then ES will be taken again to be re-examined by histology and microbiology.

ELIGIBILITY:
Inclusion criteria:

1. Age 20-45 years;
2. Women with a history of 2 or more consecutive miscarriages before 24 weeks of gestation12; or
3. Women who failed to conceive after unprotected intercourse for one year; or
4. Women who failed failure to achieve a clinical pregnancy after two consecutive cycles of IVF, ICSI or frozen embryo replacement cycles where the cumulative number of transferred embryos is no less than four for day-2 embryos and no less than 2 for day-5 embryos (blastocysts), with all embryos being of good quality.

Exclusion criteria

1. Uncorrected uterine anomalies, such as the septate or bicornuate uterus, fibroids (submucous/intramural);
2. Untreated hydrosalpinx;
3. History of antiphospholipid syndrome;
4. Known clinical autoimmune disease;
5. Undergoing immunotherapy;
6. Abnormal thyroid function;
7. Abnormal karyotyping.
8. Those with active pelvic inflammatory disease or suspicion of infection etc.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Please kindly see the inclusion criteria. The endometrics sampling is only done for female patients.
Study Population: Subjects will be identified and recruited from the IVF and miscarriage clinic by clinicians and research nurse.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 31 December 2027
  compare the brith rate between the group and cohort

SECONDARY OUTCOMES:
Compare the pregnancy rate between groups | 31 March 2028
  compare the general pregnancy rate in women with or without CE
Compare the miscarriage rate between groups | 31 March 2028
  compare the miscarriage rate in women with or without CE
Compare the implantation rate between groups | 31 March 2028
  Compare the implantation successful rate in women with or without CE

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pui Wah Chung, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No